CLINICAL TRIAL: NCT02743234
Title: Fecal Microbiota Transplantation for Relapsing Clostridium Difficile Infection
Acronym: FACIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FACIT
Record Dates: First submitted 2016-04-08; First posted 2016-04-19 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation; Fidaxomicin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FMT (Experimental): Fecal microbiota transplantation (FMT) following 4-10 days of vancomycin 125 mg x 4, using cryopreserved feces from a healthy anonymous donor
  Interventions: Other: Fecal microbiota transplantation
- Fidaxomicin (Active Comparator): 10 days fidaxomicin 200 mg x 2 daily
  Interventions: Drug: Fidaxomicin
- Vancomycin (Active Comparator): 10 days vancomycin 125 x 4 daily
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Other: Fecal microbiota transplantation — FMT follows 4-10 days of vancomycin 125 mg x 4 daily
  Arms: FMT
Drug: Fidaxomicin — Fidaxomicin 200 mg x 2 daily for 10 days
  Arms: Fidaxomicin
Drug: Vancomycin — Vancomycin 125 mg x 4 daily for 10 days
  Arms: Vancomycin

SUMMARY:
Randomized open label clinical trial to compare the clinical and microbiological efficacy of fecal microbiota transplantation, fidaxomicin, and vancomycin for relapsing Clostridium difficile infection

ELIGIBILITY:
Inclusion Criteria:

1. Relapse of Clostridium difficile infection with previous trial of vancomycin or fidaxomicin

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. Does not speak or understand the Danish language
3. Current antibiotic treatment other than metronidazole, vancomycin, fidaxomicin
4. fulminant colitis which contraindicates medical treatment
5. physician's evaluation that the patient cannot tolerate project inclusion

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with global resolution (clinical resolution AND negative Clostridium difficile PCR test) 8 weeks after primary treatment | 8 weeks
  Global resolution is defined as combined clinical and microbiological resolution, without need for rescue FMT or colectomy. Clinical resolution is absence of abdominal pain (pain score 0 (no pain), 1 (mild pain), 2 (moderate pain), 3 (severe pain)) and less than 3 bowel movements of Bristol 5 or lower, per day. Microbiological resolution is negative Clostridium difficile test 8 weeks after finishing allocated treatment

SECONDARY OUTCOMES:
Number of patients with clinical resolution 1 week after primary treatment | 1 week
  Clinical resolution (absence of abdominal pain and less than 3 bowel movements of Bristol 5 or lower, per day) 1 week after finishing allocated treatment
Number of patients with clinical resolution 8 weeks after primary treatment | 8 weeks
  Clinical resolution (absence of abdominal pain and less than 3 bowel movements of Bristol 5 or lower, per day) 8 weeks after finishing allocated treatment, without need for rescue FMT or colectomy
Number of patients with clinical resolution 26 weeks after primary treatment | 26 weeks
  Clinical resolution (absence of abdominal pain and less than 3 bowel movements of Bristol 5 or lower, per day) 26 weeks after finishing allocated treatment, without need for rescue FMT or colectomy
Number of patients with microbiological resolution week 1 | 1 week
  Microbiological resolution (negative Clostridium difficile PC test) 1 weeks after finishing allocated treatment, without need for rescue FMT or colectomy
Number of patients with microbiological resolution week 8 | 8 weeks
  Microbiological resolution (negative Clostridium difficile PC test) 8 weeks after finishing allocated treatment, without need for rescue FMT or colectomy
Number of patients with microbiological resolution week 26 | 26 weeks
  Microbiological resolution (negative Clostridium difficile PC test) 26 weeks after finishing allocated treatment, without need for rescue FMT or colectomy
Number of patients with global resolution (Clinical and microbiological resolution) week 1 | 1 week
  Clinical resolution (absence of abdominal pain and less than 3 bowel movements of Bristol 5 or lower, per day) and microbiological resolution(negative Clostridium difficile test) 1 week after finishing allocated treatment, without need for rescue FMT or colectomy
Number of patients with global resolution (Clinical and microbiological resolution) week 26 | 26 weeks
  Clinical resolution (absence of abdominal pain and less than 3 bowel movements of Bristol 5 or lower, per day) and microbiological resolution(negative Clostridium difficile test) 26 weeks after finishing allocated treatment, without need for rescue FMT or colectomy
Numerical change in quality of life (EQ5D-3L) week 8 and 26 | 8 and 26 weeks
  EQ5D-3L (www.euroqol.com) measures self-reported quality of life in 5 dimensions (each three levels), rendering score from 5 (lowest and best) to 15 (highest and worst) plus an overall reporting of general well being (0, lowest, worst to 100, highest, best). Scoring is obtained week 0,8,26 after randomization. Numerical changes are documented and compared using non-parametric statistics
Microbiota pattern changes 1, 8 and 26 weeks | 1, 8 and 26 weeks
  Microbiota profiling, 16S rRNA, absence or presence of specific genera

CONTACTS AND LOCATIONS:
Overall Officials: Jens F Dahlerup, MD DrMSc, Principal Investigator — Associate professor
Locations (1):
- Aarhus University Hospital, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hammeken LH, Baunwall SMD, Dahlerup JF, Hvas CL, Ehlers LH. Health-related quality of life in patients with recurrent Clostridioides difficile infections. Therap Adv Gastroenterol. 2022 Apr 18;15:17562848221078441. doi: 10.1177/17562848221078441. eCollection 2022. PMID 35463939
- [Derived] Hvas CL, Dahl Jorgensen SM, Jorgensen SP, Storgaard M, Lemming L, Hansen MM, Erikstrup C, Dahlerup JF. Fecal Microbiota Transplantation Is Superior to Fidaxomicin for Treatment of Recurrent Clostridium difficile Infection. Gastroenterology. 2019 Apr;156(5):1324-1332.e3. doi: 10.1053/j.gastro.2018.12.019. Epub 2019 Jan 2. PMID 30610862